CLINICAL TRIAL: NCT01055262
Title: An Open Label Study To Evaluate The Safety, Tolerability And On-Body Temperature Of A Disposable Heatwrap Device For The Lower Back
Brief Title: Safety, Tolerability And On-Body Temperature Of A Disposable Heatwrap Device For The Lower Back
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: TC-09-06; TC-09-06
Record Dates: First submitted 2010-01-21; First posted 2010-01-25 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: Safety; tolerability; heatwrap; lower back; healthy subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Heatwrap 1 (Experimental): Experimental heatwrap device for the lower back
  Interventions: Device: Heatwrap 1

INTERVENTIONS:
Device: Heatwrap 1 — 8 hours continuous topically-applied heat

SUMMARY:
The objectives of this study are to evaluate the dermal safety and on-body temperature of a disposable heatwrap product when worn while in a supine position for five consecutive days. The product will be worn on the back for approximately 8 hours per 24 hour period.

DETAILED DESCRIPTION:
Purpose-To obtain safety , tolerability and on-body temperature of a heatwrap device for the lower back.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a male or female in generally good health greater or equal to 35 years of age;
* Female subjects of child-bearing potential and those who are post-menopausal for less than 2 years must be using a medically-approved method of contraception (i.e., oral, transdermal, or implanted contraceptive hormones, cervical cap, intrauterine device, diaphragm, condom, abstinence, or surgical sterility including partner's vasectomy);
* The subject has a waist-hip circumference of between 27-47 inches inclusive.

Exclusion Criteria:

* The subject is a pregnant or lactating woman;
* The subject is diabetic;
* The subject has a history of melanoma, squamous or basal cell carcinoma in the area of application of the lower back and hip;
* The subject has any active skin disease which may contraindicate participation, including eczema, rash, broken or irritated skin, contact dermatitis and atopic dermatitis, or any skin condition that may be aggravated by heat;
* The subject has used (within the previous week) or is using any topical drug or heatwrap or electrical heat pads at the application site; or
* The subject has damaged skin in, or around the test sites which includes sunburn, uneven skin tones, tattoos, scars or other disfiguration at the application site, including an erythema grading of greater than 0 at the application site.

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2010-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=TC-09-06&StudyName=Safety%2C%20Tolerability%20And%20On-Body%20Temperature%20Of%20A%20Disposable%20Heatwrap%20Device%20For%20The%20Lower%20Back

RESULTS

PARTICIPANT FLOW:
Groups:
- ThermaCare Overnight HeatWrap: Participants wore 1 heatwrap per day for 5 consecutive days (applied to lower back, worn approximately 8 hours/day while lying in a supine position).
Period: Overall Study
Arm/Group | ThermaCare Overnight HeatWrap
Started | 169
Completed | 160
Not Completed | 9
Not completed — Adverse Event | 5
Not completed — Protocol Violation | 3
Not completed — Uncooperativeness | 1

BASELINE CHARACTERISTICS:
Arm/Group | ThermaCare Overnight HeatWrap
Number analyzed (Participants) | 169
Age Continuous [Mean (Full Range); unit: years] | 55.9 [35.0 to 87.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115
  Male | 54

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Significant Skin Event (Day 5 Cumulative)
Description: Events associated with Day X wear (eg, Day 5) assessed morning of Day X+1 (eg, Day 6). Significant skin event: at least moderate erythema, elevated response or pain upon touch (associated with non-zero erythema). Erythema grading scale: 0 (no visible erythema) to 3.0 (severe erythema, very intense redness) with 0.5 increments. Moderate erythema (2.0): definite redness. Elevated response: edema, papules, vesicle (≤ 0.5 centimeter [cm] diameter), bullae (> 0.5 cm diameter), miliaria rubra, profunda or follicular response. Pain upon touch: skin grader asked "Does your skin hurt when I touch it?"
Time Frame: Day 2 to Day 6
Population: Safety population: participants who wore the product at least once during the study
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ThermaCare Overnight HeatWrap
Number analyzed (Participants) | 169
Percentage of participants | 2.4 [0.1 to 4.7]

2. Secondary Outcome: Percentage of Participants With Significant Skin Event (Days 1 Through 4 Cumulative)
Description: Events associated with Day X wear (eg, Day 4) assessed on the morning of Day X+1 (eg, Day 5). Significant skin event: at least moderate erythema, elevated response or pain upon touch (associated with non-zero erythema). Erythema grading scale: 0 (no visible erythema) to 3.0 (severe erythema, very intense redness) with 0.5 point increments. Moderate erythema (2.0): definite redness. Elevated responses: edema, papules, vesicle (≤ 0.5 cm diameter), bullae (> 0.5 cm diameter), miliaria rubra, profunda or follicular response. Pain upon touch: skin grader asked "Does your skin hurt when I touch it?"
Time Frame: Day 2 to Day 5
Population: Safety population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ThermaCare Overnight HeatWrap
Number analyzed (Participants) | 169
Percentage of participants
  Day 1 | 1.2 [0.0 to 2.8]
  Day 2 | 1.2 [0.0 to 2.8]
  Day 3 | 2.4 [0.1 to 4.7]
  Day 4 | 2.4 [0.1 to 4.7]

3. Secondary Outcome: Time to First Significant Skin Event
Description: Significant skin event: at least moderate erythema, elevated response or pain upon touch (associated with non-zero erythema). Erythema grading scale: 0 (no visible erythema) to 3.0 (severe erythema, very intense redness) with 0.5 point increments. Moderate erythema (2.0): definite redness. Elevated responses: edema, papules, vesicle (≤ 0.5 cm diameter), bullae (> 0.5 cm diameter), miliaria rubra, profunda or follicular response. Pain upon touch: skin grader asked "Does your skin hurt when I touch it?"
Time Frame: Baseline to Day 6
Population: Safety population; Number of participants analyzed (N) = number of participants with significant skin event.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | ThermaCare Overnight HeatWrap
Number analyzed (Participants) | 4
Days | 2.0 (1.2)

4. Secondary Outcome: Percentage of Participants With Any Non-zero Erythema Score or Elevated Response (Days 1 Through 5 Cumulative)
Description: Events associated with Day X wear (eg, Day 5) assessed on the morning of Day X+1 (eg, Day 6). Erythema grading scale was a 7 point scale that ranged from 0 (no visible erythema) to 3.0 (severe erythema, very intense redness), with 0.5 point increments. Elevated responses included edema, papules, vesicle (≤ 0.5 cm diameter), bullae (> 0.5 cm diameter), miliaria rubra, profunda, or follicular response.
Time Frame: Day 2 to Day 6
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | ThermaCare Overnight HeatWrap
Number analyzed (Participants) | 169
Percentage of participants
  Day 1 | 3.0 [0.4 to 5.5]
  Day 2 | 3.6 [0.8 to 6.3]
  Day 3 | 5.3 [1.9 to 8.7]
  Day 4 | 6.5 [2.8 to 10.2]
  Day 5 | 6.5 [2.8 to 10.2]

5. Secondary Outcome: Time to First Report of Non-zero Erythema Score or Elevated Response
Description: Erythema grading scale was a 7 point scale that ranged from 0 (no visible erythema) to 3.0 (severe erythema, very intense redness), with 0.5 point increments. Elevated responses included edema, papules, vesicle (≤ 0.5 cm diameter), bullae (> 0.5 cm diameter), miliaria rubra, profunda, or follicular response.
Time Frame: Baseline to Day 6
Population: Safety population; N = participants with any application site finding
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | ThermaCare Overnight HeatWrap
Number analyzed (Participants) | 11
Days | 2.2 (1.3)

6. Secondary Outcome: Time to Worsening of Non-zero Erythema Score or Elevated Response Leading to Study Discontinuation
Description: Participants discontinued study due to adverse event (AE) if erythema ≥ 2.0, pain upon touch associated with non-zero erythema score or elevated response on the morning of Day X+1. Erythema grading scale: 0 (no visible erythema) to 3.0 (severe erythema, very intense redness) with 0.5 point increments. Elevated responses included edema, papules, vesicle (≤ 0.5 cm diameter), bullae (> 0.5 cm diameter), miliaria rubra, profunda or follicular response. Pain upon touch: skin grader asked "Does your skin hurt when I touch it?"
Time Frame: Baseline to Day 6
Population: Safety population; N = participants with a non-zero erythema score or elevated response leading to study discontinuation.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | ThermaCare Overnight HeatWrap
Number analyzed (Participants) | 4
Days | NA (NA) — Not available (NA): No participant experienced a worsening of a nonzero erythema score or elevated response leading to study discontinuation.

7. Secondary Outcome: Percentage of Participants Discontinued From Wrap Wear by 8 Hours on Any Day
Description: Skin assessments performed prior to heatwrap application; participant discontinued wrap wear for day (8 hours) if erythema score ≥ 2 with pain upon touch or elevated response. Outcome included those who discontinued wrap wear by 4 hours on same day. Erythema grading scale: 7 point scale that ranged from 0 (no visible erythema) to 3.0 (severe erythema, very intense redness) with 0.5 point increments. Moderate erythema (2.0) was definite redness. Elevated responses included edema, papules, vesicle (≤ 0.5 cm diameter), bullae (> 0.5 cm diameter), miliaria rubra, profunda or follicular response.
Time Frame: Baseline to Day 6
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | ThermaCare Overnight HeatWrap
Number analyzed (Participants) | 169
Percentage of participants | 0.6

8. Secondary Outcome: Percentage of Participants Discontinued From Wrap Wear by 4 Hours on Any Day
Description: Skin assessments performed after 4 hours of wear, participants discontinued wrap wear for remainder of day (4 hours) if erythema score ≥ 2 with pain upon touch or elevated response. Erythema grading scale: 7 point scale ranging from 0 (no visible erythema) to 3.0 (severe erythema, very intense redness) with 0.5 point increments. Moderate erythema (2.0) was definite redness. Elevated responses included edema, papules, vesicle (≤ 0.5 cm diameter), bullae (> 0.5 cm diameter), miliaria rubra, profunda and follicular response.
Time Frame: Baseline to Day 6
Population: Safety Population
Measure: Number; unit: Percentage of participants
Arm/Group | ThermaCare Overnight HeatWrap
Number analyzed (Participants) | 169
Percentage of participants | 0.6

ADVERSE EVENTS:
Arm/Group | ThermaCare Overnight HeatWrap
Serious Adverse Events (participants affected / at risk) | 0/169
Other Adverse Events (participants affected / at risk) | 10/169
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ThermaCare Overnight HeatWrap (N=169)
Application site scab (General disorders) | 5
Application site vesicles (General disorders) | 3
Application site erosion (General disorders) | 1
Application site exfoliation (General disorders) | 1
Aplication site oedema (General disorders) | 1
Application site pruritus (General disorders) | 1
Application site scar (General disorders) | 1
Skin hyperpigmentation (General disorders) | 1
Erythema (General disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.